CLINICAL TRIAL: NCT05822401
Title: Prevention, Management and Rehabilitation of Knee Osteoarthritis at the Workplace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Southern Denmark (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10429; H-22016339 (Other: Regional Scientific Ethical Committee)
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Knee Pain Chronic; Knee Osteoarthritis; Knee Discomfort
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (BFR) (Experimental): Blood flow restricted training (BFR) integrated into the daily work tasks for 8 weeks.
  Interventions: Behavioral: Blood flow restriction (BFR); Behavioral: Usual care (control)
- Usual care (control) (Active Comparator): Will continue their work as usual
  Interventions: Behavioral: Usual care (control)

INTERVENTIONS:
Behavioral: Blood flow restriction (BFR) — Blood flow restricted training integrated into the daily work tasks for 8 weeks.
  Arms: Blood flow restriction (BFR)
Behavioral: Usual care (control) — Will continue their work as usual

SUMMARY:
The goal of this intervention study is to assess the effect of blood flow restricted (BFR) exercise integrated into the daily work tasks among hospital workers with or at increased risk of chronic knee pain.

The main questions are:

Can BFR exercise integrated into the daily work tasks reduce knee pain (primary outcome) and improve function and work ability among hospital workers with or at increased risk of chronic knee pain? Participants in the intervention group will for shorts bouts during their workdays integrate BFR into their daily work tasks involving walking, whereas the control group will continue as usual.

ELIGIBILITY:
Inclusion Criteria:

* Hospital workers working at least 20 hours per week with or without chronic knee pain (>3 months)

Exclusion Criteria:

* Life-threatening disease
* Conditions where BFR training may be contraindicated, e.g. pregnancy, cancer, diabetes, major cardiovascular disease, current, previous or family history of clotting disorders, recent immobilization, major surgery or injections into the joint (i.e. corticosteroid injection)
* Systolic/diastolic blood pressure above 160/100 mmHg

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity.
Enrollment: 80 (Estimated)
Dates: Start 2023-04-11 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Change pre-post 8 weeks of intervention
  Change in worst knee pain intensity during the last week rated on a 11-point numeric rating scale (NRS)

SECONDARY OUTCOMES:
Functional performance | Change pre-post 8 weeks of intervention
  30-s chair-stand test, 40 m fast-paced walk test, a stair-climb test, maximal isometric knee extensor muscle strength
Work ability | Change pre-post 8 weeks of intervention
  Single-item on physical work ability derived from the Work Ability Index (WAI)

OTHER OUTCOMES:
Work-limiting pain | Change pre-post 8 weeks of intervention
  Rating of the degree of work limitations due to pain
Work-related fatigue | Change pre-post 8 weeks of intervention
  Rating af work-related fatigue in different body parts

IPD SHARING:
Plan to Share IPD: No